CLINICAL TRIAL: NCT07112417
Title: "A Clinical Trial Investigating the Accuracy of Augmented Reality-Guided Miniscrew Placement in Orthodontics"
Brief Title: "Augmented Reality-Assisted Miniscrew Placement in Orthodontics: A Clinical Trial"
Acronym: "AR-MSP"
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, omar hassan abd el azeem, studient of master, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AR-Ortho-MSc01
Record Dates: First submitted 2025-08-02; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-07

CONDITIONS: Orthodontic
Keywords: Augmented Reality

STUDY DESIGN:
Intervention Model Description: "This is a randomized controlled clinical trial to evaluate the effectiveness of augmented reality (AR)-guided placement of orthodontic mini-screws compared to conventional placement methods. Participants will be randomly assigned to either the AR-guided group or the conventional placement group."
Masking Description: No masking will be implemented as both participants and operators will be aware of the intervention type.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Augmented Reality-Guided Mini-Screw Placement (Active Comparator): Participants in this group will undergo mini-screw placement using augmented reality (AR) guidance to enhance accuracy and reduce placement errors
  Interventions: Device: Augmented Reality
- conventional Mini-Screw Placement (Active Comparator): Participants in this group will undergo mini-screw placement using conventional placement
  Interventions: Procedure: Conventional screw placement

INTERVENTIONS:
Device: Augmented Reality — Participants in this group will undergo mini-screw placement assisted by augmented reality (AR) technology. A customized AR system will guide the clinician in real-time to ensure optimal screw positioning, improve accuracy, and minimize placement errors.
  Arms: Augmented Reality-Guided Mini-Screw Placement
Procedure: Conventional screw placement — Participants in this group will receive mini-screw placement using the conventional freehand method without augmented reality assistance. The screws will be placed according to standard clinical protocols based on anatomical landmarks and clinician experience
  Arms: conventional Mini-Screw Placement

SUMMARY:
This study aims to evaluate the effectiveness and accuracy of using Augmented Reality (AR) technology in the placement of mini-screws (Temporary Anchorage Devices) during orthodontic treatment. By combining CBCT images with digital dental scans and visualizing them using AR, clinicians can place mini-screws more precisely. The study is a pilot clinical trial involving patients at the Faculty of Dentistry, Al-Azhar University - Assiut Branch.

DETAILED DESCRIPTION:
This is a pilot clinical trial designed to assess the feasibility and accuracy of augmented reality (AR)-guided mini-screw insertion in orthodontic patients. The study involves the use of CBCT imaging and digital intraoral scanning to create a 3D model of the patient's jaw. This model is then processed and integrated into an AR platform that allows real-time visualization of the ideal screw insertion site.

Participants are selected based on inclusion and exclusion criteria. After obtaining informed consent, CBCT and intraoral scans are performed. The proposed mini-screw location is determined digitally and projected using an AR device (tablet or headset) during the clinical procedure.

After insertion, a follow-up CBCT scan is taken to evaluate the deviation between the planned and actual screw positions (linear and angular deviation). Data on insertion time, patient comfort, and operator satisfaction will also be recorded.

The study is conducted at the Faculty of Dentistry, Al-Azhar University - Assiut Branch, with prior ethical approval obtained from the institutional review board.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients indicated for orthodontic mini-screw placement as part of their treatment plan.

  2. Age between 15 and 40 years.

  3. Good general health (ASA I or II).

  4. Adequate oral hygiene and healthy periodontal condition.

  5. Ability to understand and provide informed consent (or guardian consent for minors).

Exclusion Criteria:

* 1 . Systemic conditions affecting bone healing (e.g., uncontrolled diabetes, osteoporosis).

  2. History of craniofacial trauma, surgery, or congenital anomalies in the maxillofacial region.

  3. Ongoing periodontal disease or poor oral hygiene.

  4. Pregnancy or lactation.

  5. Use of medications influencing bone metabolism (e.g., bisphosphonates, corticosteroids).

  6. Allergy to local anesthetics or materials used in the procedure.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-08-31 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy of screw placement | 1 week post-op
  Accuracy will be assessed using CBCT imaging compared to planned position

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No
NO plan to share